CLINICAL TRIAL: NCT00897208
Title: Estrogen-DNA Adducts in Breast, Urine and Serum as Biomarkers of Breast Cancer Risk
Brief Title: Studying Biomarkers in Nipple Fluid, Urine, and Blood Samples From Women With Newly Diagnosed Ductal Carcinoma In Situ or Stage I or Stage II Breast Cancer and in Women at Risk of Developing Breast Cancer
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 19-2005; 19-2005 (Other: Mayo Clinic Cancer Center); 06-008665 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Breast Cancer
Keywords: breast cancer; ductal breast carcinoma in situ; breast cancer in situ; stage IA breast cancer; stage IB breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ | interventions — Chromatography, High Pressure Liquid; Mass Spectrometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: high performance liquid chromatography
Other: laboratory biomarker analysis
Other: mass spectrometry
Other: medical chart review
Procedure: evaluation of cancer risk factors

SUMMARY:
RATIONALE: Studying samples of nipple fluid, urine, and blood in the laboratory from patients with cancer and from patients at risk of developing cancer may help doctors identify and learn more about biomarkers related to cancer. It may also help doctors learn more about breast cancer and identify patients at risk of developing breast cancer.

PURPOSE: This laboratory study is looking at biomarkers in nipple fluid, urine, and blood samples from women with newly diagnosed ductal carcinoma in situ or stage I or stage II breast cancer and in women at risk of developing breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the levels of catechol estrogens (CE), CE metabolites, CE-DNA adducts, and CE conjugates in nipple aspirate fluid samples obtained from women with newly diagnosed ductal carcinoma in situ or stage I or II breast cancer and from women at high risk of developing breast cancer.

OUTLINE: Patients with newly diagnosed breast cancer or at high risk of developing breast cancer undergo nipple aspiration. The nipple aspirate fluid is obtained from the unaffected breast and is analyzed for 31 estrogen metabolites, conjugates, and depurinating DNA adducts by high-performance liquid chromatography (LC) with electrochemical and mass spectrometric detectors. All patients undergo urine and serum sample collection. The urine samples are analyzed by ultraperformance LC monitored by tandem mass spectrometry for estrogen metabolites, conjugates, and depurinating DNA adducts.

Patients' charts are reviewed to obtain information about age, race, general health, any endocrine disorders, history of cancer, estrogen and progesterone receptor status, and HER2/neu status (for patients with newly diagnosed breast cancer), menopausal status, reproductive history, history of breast disease, medication use, smoking history, and history of alcohol consumption.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Newly diagnosed (within 30 calendar days of diagnosis) stage I or II breast cancer

    * Node-negative or node-positive disease
  * Newly diagnosed ductal carcinoma in situ (stage 0) of the breast
  * At high risk of developing breast cancer, as indicated by at least 1 of the following criteria:

    * Gail model 5-year risk score ≥ 1.66%
    * Gail model lifetime-risk estimate ≥ 20%
    * Known deleterious BRCA 1 or 2 gene mutation carrier
    * History of lobular carcinoma in situ or atypical ductal or lobular hyperplasia
  * At low or average risk of developing breast cancer (control group)

    * Gail model 5-year risk score < 1.66% or lifetime risk < 20%
* No advanced breast cancer
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Pre- or post-menopausal

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for breast cancer or any other cancer
* More than 3 months since prior and no concurrent estrogen or other hormones
* More than 3 months since prior oral contraceptives
* No concurrent selective estrogen receptor modulators (tamoxifen citrate or raloxifene)
* No concurrent aromatase inhibitors

Ages: 19 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population is adult women, ages 19 to 80 years of age. In 2003, there were approximately 2000 new and 3000 established patient visits in the Breast Diagnostic Clinic (BDC) and Breast Cancer Clinic (BCC) Our new patients include those seen in the BDC with new breast concerns and those at seeking counseling regarding a family history or at high risk for developing breast cancer, as well as those women seen in the BCC with a new diagnosis of invasive or non-invasive breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2005-05-20 (Actual); Primary Completion 2010-06-17 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Comparison of the levels of estrogens, catechol estrogen (CE) metabolites, CE-glutathione conjugates, and CE-DNA adducts (N3Ade and N7Gua) among healthy women, high-risk women, and women with breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Sandhya Pruthi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Cancer Center, Rochester, Minnesota, United States